CLINICAL TRIAL: NCT06793943
Title: A Phase 1, Open-Label, 4-Part Trial to Assess the Drug-Drug Interaction Between Zasocitinib and Combined Oral Contraceptives, a MATE Substrate, a P-gp Substrate, and a Proton-Pump Inhibitor in Healthy Participants
Brief Title: A Study of Interaction of Zasocitinib (TAK-279) With Other Medicines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-279-1011
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — Metformin; Digoxin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: COC (LNG and EE) + Zasocitinib (Experimental)
  Interventions: Drug: Zasocitinib; Drug: COC
- Part 2: Metformin + Zasocitinib (Experimental)
  Interventions: Drug: Zasocitinib; Drug: Metformin
- Part 3: Digoxin + Zasocitinib (Experimental)
  Interventions: Drug: Zasocitinib; Drug: Digoxin
- Part 4: Zasocitinib + Esomeprazole (Experimental)
  Interventions: Drug: Zasocitinib; Drug: Esomeprazole

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib tablets specified doses on specified days.
  Other Names: TAK- 279
Drug: COC — COC tablets (containing LNG and EE) specified doses on specified days.
  Arms: Part 1: COC (LNG and EE) + Zasocitinib
Drug: Metformin — Metformin tablets specified doses on specified days.
  Arms: Part 2: Metformin + Zasocitinib
Drug: Digoxin — Digoxin tablets specified doses on specified days.
  Arms: Part 3: Digoxin + Zasocitinib
Drug: Esomeprazole — Esomeprazole capsules specified doses on specified days.
  Arms: Part 4: Zasocitinib + Esomeprazole

SUMMARY:
The main aim of this study is to find out how zasocitinib (TAK-279) interacts with other medicines taken by mouth (orally). This will be examined by how the body processes medicines, which is called pharmacokinetics or PK. In this study, other medicines that will be administered together with zasocitinib include a contraceptive (levonorgestrel (LNG) and ethinyl estradiol [EE]), a medicine for diabetes (metformin), a medicine used for heart problems (digoxin), and a medicine that blocks the production of stomach acid (esomeprazole).

Another aim is to learn about the side effects of zasocitinib and how well it is tolerated when taken alone and together with these other medicines.

During the study, participants will need to stay at the clinic for up to 27 days.

DETAILED DESCRIPTION:
The drug being tested in this study is called zasocitinib.

Zasocitinib is being tested to assess the effect of zasocitinib on the pharmacokinetics of Combined Oral Contraceptive (COC [containing LNG and EE] in Part 1), multidrug and toxic compound extrusion (MATE) substrate (metformin in Part 2), and a P-glycoprotein (P-gp) substrate (digoxin in Part 3). Additionally, the effect of proton-pump inhibitor (PPI) (esomeprazole in Part 4) on the pharmacokinetics of zasocitinib is being evaluated in healthy participants.

The study will enroll approximately 78 participants. Participants will be enrolled in one of the four parts to evaluate the following treatments:

* Part 1: COC (LNG and EE) + Zasocitinib
* Part 2: Metformin + Zasocitinib
* Part 3: Digoxin + Zasocitinib
* Part 4: Zasocitinib + Esomeprazole

The overall time (including screening and follow-up periods) to participate is approximately 68 days for Part 1, 54 days for Part 2, 62 days for Part 3 and 56 days for Part 4. All participants will be followed up for up to 14 days after the last dose of Period 2 in each Part.

ELIGIBILITY:
Inclusion criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilograms per square meter (kg/m^2) at the screening visit.
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and Electrocardiograms (ECGs) as outlined in the protocol.

   Part 1 Only:
3. Healthy, adult, female, aged 18 to 65 years, inclusive, at the screening visit.

   Parts 2-4 Only:
4. Healthy, adult, male or female, aged 18 to 55 years, inclusive, at the screening visit.

Exclusion criteria:

1. Positive urine drug or alcohol results at the screening visit or at check-in.
2. Unable to refrain from or anticipates the use of:

   * Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements and other drugs outlined in protocol.
   * Any drugs known to be inducers of Cytochrome P450 3A4 (CYP3A4) and/or P-gp, including St. John's Wort, for 28 days prior to the first dosing.
3. Has been on a diet incompatible with the on-trial diet, in the opinion of the investigator or designee, within the 30 days prior to first dosing and throughout the trial.
4. Has made a donation of blood or had significant blood loss within 56 days prior to first dosing.
5. Has made a plasma donation within 7 days prior to first dosing.
6. Participated in another clinical trial within 30 days prior to first dosing. The 30-day window will be derived from the date of the last dosing in the previous trial to Day 1 of Period 1 of the current trial.
7. Has herpes infections.
8. Positive results for non-herpetic viral diseases at the screening visit.
9. Positive results for tuberculosis (TB) at the screening visit.

   Part 1:
10. Unable to refrain from or anticipates the use of:

    * Any drugs known to increase or decrease levels of sex hormone-binding globulin (SHBG), including any oral, topical, or intravaginal hormone-containing product, within 12 weeks prior to the first dosing.
    * Any injectable or implantable hormone-containing product within 1 year prior to the first dosing.

    Part 2 Only:
11. Hemoglobin A1c (HbA1c) greater than (>) ULN (5.7 percentage [%]) and deemed clinically significant by the investigator or designee at the screening visit.

    Part 3 Only:
12. Has or is at risk for major cardiac events or dysfunction.

    Part 4 Only:
13. Had diarrhea or vomiting within 48 hours prior to check-in.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Part 1: Cmax: Maximum Observed Plasma Concentration for LNG and EE When Administered Alone and With Zasocitinib | Up to 144 hours
Part 1: AUCinf: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for LNG and EE When Administered Alone and With Zasocitinib | Up to 144 hours
Part 1: AUClast: Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration for LNG and EE When Administered Alone and With Zasocitinib | Up to 144 hours
Part 2: Cmax for Metformin When Administered Alone and With Zasocitinib | Up to 48 hours
Part 2: AUCinf for Metformin When Administered Alone and With Zasocitinib | Up to 48 hours
Part 2: AUClast for Metformin When Administered Alone and With Zasocitinib | Up to 48 hours
Part 3: Cmax for Digoxin When Administered Alone and With Zasocitinib | Up to 144 hours
Part 3: AUCinf for Digoxin When Administered Alone and With Zasocitinib | Up to 144 hours
Part 3: AUClast for Digoxin When Administered Alone and With Zasocitinib | Up to 144 hours
Part 4: Cmax for Zasocitinib When Administered Alone and With Esomeprazole | Up to 120 hours
Part 4: AUCinf for Zasocitinib When Administered Alone and With Esomeprazole | Up to 120 hours
Part 4: AUClast for Zasocitinib When Administered Alone and With Esomeprazole | Up to 120 hours

SECONDARY OUTCOMES:
Parts 1, 2, 3 and 4: Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESIs) | Part 1: Up to 33 days; Part 2: Up to 23 days; Part 3: Up to 27 days; Part 4: Up to 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/b330809145414f2b??page=1&idFilter=TAK-279-1011